CLINICAL TRIAL: NCT01807403
Title: Comparison of the Efficacy of Subthalamic Nucleus, Caudate Nucleus and Nucleus Accumbens Electric Stimulation in Severe and Resistant Obsessive-compulsive Disorder.
Brief Title: Comparison of DBS Targets in Obsessive-compulsive Disorder
Acronym: PRESTOC2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P081203
Record Dates: First submitted 2013-01-25; First posted 2013-03-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Deep brain stimulation; Subthalamic nucleus; Caudate nucleus; Nucleus accumbens
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Deep brain stimulation of subthalamic nucleus (Experimental): Pose of bilateral subthalamic and caudate stimulating macroelectrodes with subclavicular pacemaker.Stimulation of subthalamic nucleus
  Interventions: Procedure: Deep brain stimulation
- Deep brain stimulation of caudate nucleus (Experimental): Pose of bilateral subthalamic and caudate stimulating macroelectrodes with subclavicular pacemaker. Caudate nucleus stimulation
  Interventions: Procedure: Deep brain stimulation
- Deep brain stimulation of nucleus accumbens (Experimental): Pose of bilateral subthalamic and caudate stimulating macroelectrodes with subclavicular pacemaker.Nucleus accumbens stimulation.
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — Pose of bilateral subthalamic and caudate stimulating macroelectrodes with subclavicular pacemaker.

SUMMARY:
Deep brain stimulation (DBS) has been proposed for severe and resistant obsessive-compulsive disorder. This electrical stimulation has been tested on, and shown to be effective at, different targets (subthalamic nucleus, caudate nucleus & nucleus accumbens). However, the efficacies of each target have never been compared directly.

This protocol aims to do so, with the hypothesis that subthalamic (STN) stimulation will be more efficacious.

DETAILED DESCRIPTION:
Deep brain stimulation has been proposed for severe and resistant obsessive-compulsive disorder (OCD). This electrical stimulation has been tested on, and shown to be effective at, different targets (subthalamic nucleus, caudate nucleus & nucleus accumbens). However, the efficacies of each target have never been compared directly.

Therefore, bilateral subthalamic and caudate electrodes will be implanted in severe OCD patients. Efficacy of stimulation at the different targets will be assessed using a double-blind randomised crossover design.

ELIGIBILITY:
Inclusion criteria :

* Age 18 - 60
* OCD according to DSM IV, at least 5 years since diagnosis
* Severe OCD responsible for a clinically significant and objective alteration of psychosocial functioning and suffering: YBOCS score>25, CGI score >= 4 and EGF score <= 40
* Resistance of OCD to at least 3 antidepressants from the serotonin reuptake inhibitors category, including clomipramine, given for at least 12 weeks with doses of at least 80mg/d for fluoxetine, 300mg/d for fluvoxamine, 200mg/d for sertraline, 60mg/d for paroxetine and citalopram, 250mg/d for clomipramine). Plus resistance to each of these 3 antidepressant associated first to risperidone or pimozide for a month then to Lithium carbonate, clonazepam, buspirone or pindolol for a month
* Resistance to at least 2 behavioural and cognitive therapies conducted by as many different specialists, following validated protocols (e.g. exposition and prevention of response)
* Oral and written knowledge of French
* Social security coverage
* Written consent of the patient after clear description of the study

Exclusion criteria :

* cognitive alteration with PM38 score < IQ85
* Other axis 1 disorder according to DSM IV, excepted, global anxiety disorder, social phobia, nicotine dependance, and antecedent of major depressive episodes
* suicidal risk >=2 on item 10 of MADRS (Montgomery Asberg Depression Rating Scale)
* Personality disorder (axis 2 of DSM IV assessed using the SCID II)
* Contra indication to MRI, abnormal brain MRI, other severe intercurrent disease
* Fertile woman without adequate contraception
* Pregnancy
* Forced psychiatric hospitalisation
* Any kind of legal protection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Severity of symptoms after each phase | 3 months
  Severity as measured by the Yale-Brown Obsession and Compulsion scale

SECONDARY OUTCOMES:
Severity of symptoms after each phase | month 0
  Severity as measured by the Yale-Brown Obsession and Compulsion scale
Severity of symptoms after each phase | 6 months
  Severity as measured by the Yale-Brown Obsession and Compulsion scale
Severity of symptoms after each phase | 10 months
  Severity as measured by the Yale-Brown Obsession and Compulsion scale
Severity of symptoms after each phase | 14 months
  Severity as measured by the Yale-Brown Obsession and Compulsion scale

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mallet, MD, PhD, Principal Investigator — Assitance Publique - Hopitaux de Paris
Locations (1):
- Centre d'investigation Clinique Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No